CLINICAL TRIAL: NCT05526365
Title: Impact of Reduced Idea Density on Pharmacy Students' Attainment in Pharmaceutical Calculations: a Single-blind Multicentre Randomised Controlled Trial
Brief Title: Idea Density in Exam Performance
Acronym: IDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: University of Central Lancashire (Other); Aston University (Other); University of Birmingham (Other); University of Bradford (Other); De Montfort University (Other); University of Greenwich (Other); University of Huddersfield (Other); Kingston University (Other); Newcastle University (Other); Queen's University, Belfast (Other); Robert Gordon University (Other); University of Ulster (Other); University of Wolverhampton (Other)
Responsible Party: Principal Investigator, Andrew Lunn, Lecturer in Clinical Pharmacy, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 22/PBS/004
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Medical Education; Health Education; Educational Assessment
Keywords: Pedagogy; Medical education; Assessment; Linguistics; Idea density
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: Participants randomised to two arms, control and intervention
Who Masked: Participant
Masking Description: Students will be blinded to allocation; performed using sequentially generated random numbers. The control and intervention exams will be identical in all but the idea density of the questions.
  The students are the unit of randomisation and intervention. As the randomisation will be 1:1, the block size multiplier will be 2, 4, 6 and the block size 4, 8, and 12. This approach will reduce bias and balance allocating participants to the treatment arm. Furthermore, the process will adopt block permutation, meaning that treatment assignments within blocks are determined to be random in order but that the desired allocation proportions are achieved exactly within each block.
  A computerised random number generator will generate the sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will receive an initial 12 question baseline test (same as intervention). They will after two weeks receive a second test that is linguistically the same as the national GPhC exam.
- Intervention (Experimental): Participants in the intervention group will receive an initial 12 question baseline test (same as control). They will after two weeks receive a second test that is reduced in idea density by around 10% overall.
  Interventions: Other: Reduced Idea Density

INTERVENTIONS:
Other: Reduced Idea Density — Question idea density reduced (ratio of propositions to total words used).
  Arms: Intervention

SUMMARY:
Text can be written in multiple ways to mean the same thing; changing how a text is written can make it easier or harder to understand. How many concepts or ideas there are in a text, divided by the total number of words, is one possible way to determine how easy or hard it is to understand. This ratio is called idea density (ID).

Varying ID has been shown to affect the speed at which a reader understands; it impacts certain people more than others, such as second language speakers. This effect may be of particular importance in an exam, where understanding a question in a limited time is key. In the UK, pharmacy students must undertake an exam set by the General Pharmaceutical Council (GPhC) to be registered as pharmacists. The exam involves pharmaceutical calculations and shows variable pass rates. This study aims to evaluate the impact of reducing ID in a pharmaceutical calculation test and will be conducted in 14 schools of pharmacy in the UK. All participants will take a GPhC style test. Then, participants will be divided into two groups of equal size; one group will undertake a second test with the same ID as the first, while the second group will undertake a test with a lower ID. Finally, the investigators will compare the second test scores between the two groups as cohorts and question by question, evaluating whether lowering ID has increased students' scores.

If and effect is seen, ensuring that questions are written with a controlled ID may help ensure we are examining more fairly and allowing students with the requisite knowledge to pass.

DETAILED DESCRIPTION:
Pharmaceutical Council must be undertaken. It involves pharmaceutical calculations and shows variable pass rates. Linguistic factors, such as idea density, affect and predict comprehension time. This trial will evaluate the effect of lowering question idea density on attainment in a pharmaceutical calculations exam aligned to that of the General Pharmaceutical Council.

Methods: This is a single-blind, parallel 2-arm multicentre randomised controlled trial conducted in fourteen Universities across the United Kingdom. A 1:1 randomisation and a sample size of 188 pharmacy students will be sufficient to detect a 1-point difference in the mean scores between the intervention and control group during a pharmacy calculation test with two-tails, 80% power and 5% significance level. Each school will recruit a minimum of 14/15 students. Participants will sit two 12-question pharmaceutical calculation tests. All participants will take the same baseline test; then, will be randomised and undertake a second test 2-week after, with standard idea density for the control group and lower idea density for the intervention. Primary outcome: the scores obtained by the participants undertaking the second calculation test 2-week after the baseline. Secondary outcomes: percentage of students achieving a pass during the second test; effect of demographic characteristics (first or not-first English language speakers, age, ethnicity, year of study, specific learning disability) on participants' attainment when lowering idea density.

Conclusion: Results could inform the development of new standards in the pharmaceutical calculations exam.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Registered as a student on an MPharm course in the UK
* Be in years 1-4 of the course (levels 1-7)

Exclusion Criteria:

* Under 18
* Not registered on an MPharm course in the UK
* Are currently undertaking a foundation year (level 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Overall performance on test 2 | 1 month
  The primary outcome is the performance in the second calculation test 2. Overall score per student can be between 0-12, and performance of all students on each question a decimal percent between 0-1, with 0 meaning 0% of students answered correctly and 1 meaning 100% of students answered correctly.

SECONDARY OUTCOMES:
Pass rate | 1 month
  The percentage of students achieving a pass (equivalent to 70% or above) during the second test.
Demographic | 1 month
  The effect of each demographic characteristic on students' attainment in pharmacy calculation when lowering idea density?
  * First language speaker (English as the first language) or not
  * Age
  * Ethnicity
  * Year of study
  * Specific learning disability

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study protocol to be published Original (anonymised) data to be placed on university repository
Supporting Information: Study Protocol
Time Frame: Within 1 year of study (when published), indefinitely available on university repository